CLINICAL TRIAL: NCT03771339
Title: Comparison of Ultrasound-Guided Quadratus Lumborum Block and Epidural Analgesia for Postoperative Pain Management After Renal Transplantation
Brief Title: Comparison of Quadratus Lumborum Block and Epidural Analgesia Following Kidney Transplant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal investigator, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes030
Record Dates: First submitted 2018-12-06; First posted 2018-12-11 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
Keywords: quadratus lumborum block; continuous epidural; postoperative analgesia; kidney transplant
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Epidural Analgesia (Active Comparator): Continuous epidural analgesia using ropivacaine 0.375% 3 mL boluses followed by ropivacaine 0.2% with rate 6 mL per hour for 24 hours
  Interventions: Procedure: Continuous Epidural analgesia
- Bilateral Quadratus Lumborum Block (Experimental): Bilateral Quadratus lumborum block using ropivacaine 0.2% 20 mL each injection after surgery
  Interventions: Procedure: Bilateral Quadratus Lumborum block

INTERVENTIONS:
Procedure: Continuous Epidural analgesia — Continuous Epidural catheter is inserted at the Thoracic 11-T12 level, using Ropivacaine 0.375% 3 mL bolus followed by Ropivacaine 0.2% with rate 6 mL/hour for 24 hours after laparoscopic nephrectomy
  Arms: Continuous Epidural Analgesia
Procedure: Bilateral Quadratus Lumborum block — Bilateral anterior Quadratus Lumborum block using Ropivacaine 0.375% 20 mL each injection as postoperative analgesia treatment for 24 hours
  Arms: Bilateral Quadratus Lumborum Block

SUMMARY:
Quadratus lumborum block as an alternative for postoperative analgesia compared with epidural block

DETAILED DESCRIPTION:
Epidural analgesia is the main choice of analgesia following kidney transplant surgery. However, continuous epidural technique had some concerning side effects such as hemodynamic instabilities, urine retention, motor/sensory disturbances/weakness, and mobilisation comfort, it could also cause hypotension which could affect graft success. Quadratus lumborum (QL) block had lesser side effects thus could be an option for postoperative analgesia, however there are no study showing the safety and success rate of QL block techniques for patients who underwent kidney transplant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective kidney transplant laparotomy surgery
* Agrees to participate in research
* BMI < 30 kg/m2

Exclusion Criteria:

* Declines to participate in research
* Contraindications to intervention procedures (epidural or quadratus lumborum block)
* History of local anaesthetic allergy
* Systemic allergic reactions, anaphylactic reaction, cardiac arrest
* Failure of intervention procedures (epidural or quadratus lumborum block)
* Intraoperative complications (massive bleeding, hypotension)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours
  Additional analgesia required at 2, 6, 12, and 24 hours after surgery

SECONDARY OUTCOMES:
Pain Intensity | 24 hours
  Pain intensity measured using the Visual Analogue Scale (VAS) at 2, 6, 12, and 24 hours after surgery. VAS assessed with horizontal line 0-100 mm for no pain to the worst pain, with range 0-30 mm for none to mild pain, 31-70 mm for moderate pain, 71-100 mm for severe pain.
First time morphine required | 24 hours
  Total time gap from postoperative analgesia procedure administration to first morphine requirement
Total minimum and maximum dose of vasoactive agents | 24 hours
  Minimum and maximum dose of norepinephrine and dobutamine as vasoactive agents within 24 hours after surgery
Urine output | 24 hours
  Urine output (mL/kgBW/hour) after surgery
Bromage score | 24 hours
  Bromage score at 2, 6, 12, and 24 hours after surgery to assess lower limb motoric block.
  Score for Bromage:
  1. free movement
  2. partial block
  3. almost complete
  4. complete block
Ramsay score | 24 hours
  Ramsay score at 2, 6, 12, and 24 hours after surgery to assess patient sedation level.
Dermatomal coverage of analgesia procedure | Immediately after anaesthesia completion
  dermatome sensory block distribution using cold sensation test
Blood ropivacaine level | 24 hours
  Arterial blood sample of all subjects will be withdrawn approximately 3 mL from the arterial line at 0, 30, 45, 60 minute, and 2, 4, 6,12,18, 24 hours after designated analgesia procedure, and will be used for ropivacaine blood level measurements using High-Performance Liquid Chromatography (HPLC), to measure Total plasma ropivacaine concentration (Cstop), maximum plasma concentration (Cmax), time of maximum plasma concentration, area under the curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, M.D., Principal Investigator — Indonesia University
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mochtar CA, Alfarissi F, Soeroto AA, Hamid ARAH, Wahyudi I, Marbun MBH, et al. Milestones of kidney transplantation in Indonesia. Med J Indones. 2017 Nov 27;26(3):229.
- [Background] Kakaei F, Nikeghbalian S, Ali S. Kidney Transplantation Techniques. In: Rath T, editor. Current Issues and Future Direction in Kidney Transplantation [Internet]. InTech; 2013 [cited 2018 Jun 6]. Available from: http://www.intechopen.com/books/current-issues-and-future-direction-in-kidney-transplantation/kidney-transplantation-techniques
- [Background] Pham PC, Khaing K, Sievers TM, Pham PM, Miller JM, Pham SV, Pham PA, Pham PT. 2017 update on pain management in patients with chronic kidney disease. Clin Kidney J. 2017 Oct;10(5):688-697. doi: 10.1093/ckj/sfx080. Epub 2017 Aug 18. PMID 28979781
- [Background] Abdelsalam K., Sultan S. Effectiveness of ultrasound-guided transversus abdominis plane block for intraoperative and postoperative analgesia in kidney transplantation. Ain-Shams J Anaesthesiol. 2015;8(1):140.
- [Background] Srivastava D, Tiwari T, Sahu S, Chandra A, Dhiraaj S. Anaesthetic management of renal transplant surgery in patients of dilated cardiomyopathy with ejection fraction less than 40%. Anesthesiol Res Pract. 2014;2014:525969. doi: 10.1155/2014/525969. Epub 2014 Aug 19. PMID 25210514
- [Background] S Martinez B. Anesthesia for Kidney Transplantation-A Review. J Anesth Clin Res [Internet]. 2013 [cited 2018 Jun 6];04(01). Available from: https://www.omicsonline.org/anesthesia-for-kidney-transplantation-a-review-2155-6148.1000270.php?aid=11555
- [Background] Hirata ES, Baghin MF, Pereira RI, Alves Filho G, Udelsmann A. Influence of the anesthetic technique on the hemodynamic changes in renal transplantation: a retrospective study. Rev Bras Anestesiol. 2009 Mar-Apr;59(2):166-76. doi: 10.1590/s0034-70942009000200004. English, Portuguese. PMID 19488528
- [Background] Aulakh NK, Garg K, Bose A, Aulakh BS, Chahal HS, Aulakh GS. Influence of hemodynamics and intra-operative hydration on biochemical outcome of renal transplant recipients. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):174-9. doi: 10.4103/0970-9185.155144. PMID 25948896
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Krohg A, Ullensvang K, Rosseland LA, Langesaeter E, Sauter AR. The Analgesic Effect of Ultrasound-Guided Quadratus Lumborum Block After Cesarean Delivery: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):559-565. doi: 10.1213/ANE.0000000000002648. PMID 29135590
- [Background] Mieszkowski MM, Mayzner-Zawadzka E, Tuyakov B, Mieszkowska M, Zukowski M, Wasniewski T, Onichimowski D. Evaluation of the effectiveness of the Quadratus Lumborum Block type I using ropivacaine in postoperative analgesia after a cesarean section - a controlled clinical study. Ginekol Pol. 2018;89(2):89-96. doi: 10.5603/GP.a2018.0015. PMID 29512813
- [Background] Lemmens HJ. Kidney transplantation: recent developments and recommendations for anesthetic management. Anesthesiol Clin North Am. 2004 Dec;22(4):651-62. doi: 10.1016/j.atc.2004.05.007. PMID 15541928
- [Background] Hockett MM, Hembrador S, Lee A. Continuous Quadratus Lumborum Block for Postoperative Pain in Total Hip Arthroplasty: A Case Report. A A Case Rep. 2016 Sep 15;7(6):129-31. doi: 10.1213/XAA.0000000000000363. PMID 27513972
- [Background] Mukhtar K, Khattak I. Transversus abdominis plane block for renal transplant recipients. Br J Anaesth. 2010 May;104(5):663-4. doi: 10.1093/bja/aeq077. No abstract available. PMID 20400617
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Schmid S, Jungwirth B. Anaesthesia for renal transplant surgery: an update. Eur J Anaesthesiol. 2012 Dec;29(12):552-8. doi: 10.1097/EJA.0b013e32835925fc. PMID 23010898
- [Background] Williams M, Milner QJ. Postoperative analgesia following renal transplantation - current practice in the UK. Anaesthesia. 2003 Jul;58(7):712-3. doi: 10.1046/j.1365-2044.2003.32661.x. No abstract available. PMID 12790818
- [Background] Nair A. Bilateral quadratus lumborum block for post-caesarean analgesia. Indian J Anaesth. 2017 Apr;61(4):362-363. doi: 10.4103/ija.IJA_204_17. No abstract available. PMID 28515533
- [Background] Ashok J, Mayur M, Asit K P, Neelam S.Postoperative Analgesia by Transmuscular Quadratus Lumborum Block Catheters. J Anest & Inten Care Med. 2016; 1(3) : 555562
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Carline L, McLeod GA, Lamb C. A cadaver study comparing spread of dye and nerve involvement after three different quadratus lumborum blocks. Br J Anaesth. 2016 Sep;117(3):387-94. doi: 10.1093/bja/aew224. PMID 27543534
- [Background] Elsharkawy H. Quadratus Lumborum Blocks. Adv Anesth. 2017;35(1):145-157. doi: 10.1016/j.aan.2017.07.007. Epub 2017 Oct 3. No abstract available. PMID 29103570
- [Background] Garg C, Khanna S, Mehta Y. Quadratus lumborum block for post-operative pain relief in patient with Prune belly syndrome. Indian J Anaesth. 2017 Oct;61(10):840-842. doi: 10.4103/ija.IJA_246_17. PMID 29242658
- [Background] Shaaban M, Esa WA, Maheshwari K, Elsharkawy H, Soliman LM. Bilateral Continuous Quadratus Lumborum Block for Acute Postoperative Abdominal Pain as a Rescue After Opioid-Induced Respiratory Depression. A A Case Rep. 2015 Oct 1;5(7):107-11. doi: 10.1213/XAA.0000000000000188. PMID 26402020
- [Background] Akerman M, Pejcic N, Velickovic I. A Review of the Quadratus Lumborum Block and ERAS. Front Med (Lausanne). 2018 Feb 26;5:44. doi: 10.3389/fmed.2018.00044. eCollection 2018. PMID 29536008
- [Background] Agrawal P, Farag E. Ultrasound-guided quadratus lumborum and subcostal transversus abdominis plane blocks. Tech Reg Anesth Pain Manag. 2014 Oct;18(4):163-5
- [Background] Brull R, MacFarlane AJR, Chan VWS. Spinal, Epidural, and Caudal Anesthesia. In: Miller RD, Cohen NH, Eriksson LI, Fleisher LA, Wiener-Kronish JP, Young WL, editors. Miller's anesthesia. Eighth edition. Philadelphia, PA: Elsevier/Saunders; 2015. p. 1684-720
- [Background] Butterworth JF, Mackey DC, Wasnick JD, Morgan GE, Mikhail MS, Morgan GE. Spinal, Epidural, & Caudal Blocks. In: Morgan and Mikhail's clinical anesthesiology. 5th ed. McGraw-Hill; 2013. p. 937-74
- [Background] Clemente A, Carli F. The physiological effects of thoracic epidural anesthesia and analgesia on the cardiovascular, respiratory and gastrointestinal systems. Minerva Anestesiol. 2008 Oct;74(10):549-63. PMID 18854796
- [Background] Wheatley RG, Schug SA, Watson D. Safety and efficacy of postoperative epidural analgesia. Br J Anaesth. 2001 Jul;87(1):47-61. doi: 10.1093/bja/87.1.47. No abstract available. PMID 11460813
- [Background] Grass JA. Patient-controlled analgesia. Anesth Analg. 2005 Nov;101(5 Suppl):S44-S61. doi: 10.1213/01.ANE.0000177102.11682.20. PMID 16334492
- [Background] Francesca F, Bader P, Echtle D, Giunta F, Williams J; EAU. EAU guidelines on pain management. Eur Urol. 2003 Oct;44(4):383-9. doi: 10.1016/s0302-2838(03)00321-x. PMID 14499670